CLINICAL TRIAL: NCT00768911
Title: Phase 1, Open Label, Multi-Center Study To Evaluate The Safety And Tolerability of CT-322 Administered In Combination With Focal Brain Radiotherapy And Temozolomide To Subjects With Newly Diagnosed Glioblastoma Multiforme
Brief Title: CT-322 in Combination With Radiation Therapy and Temozolomide to Treat Newly Diagnosed Glioblastoma Multiforme
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adnexus, A Bristol-Myers Squibb R&D Company (Industry)
Responsible Party: Medical Director, Adnexus, A Bristol-Myers Squibb R&D Company, Adnexus, A Bristol-Myers Squibb R&D Company
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-322.003
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-10

CONDITIONS: Glioblastoma Multiforme
Keywords: glioblastoma; Glioblastoma multiforme (newly diagnosed)
MeSH Terms: conditions — Glioblastoma | interventions — CT-322; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: CT-322; Drug: Temozolomide; Procedure: Radiation Therapy

INTERVENTIONS:
Drug: CT-322 — Intravenous solution, intravenous administration, starting dose level of 0.5 mg/kg/week
  Dose levels: 0.5 mg/kg/week, 1.0 mg/kg/week, 2.0 mg/kg/week
Drug: Temozolomide — 75 mg/M2/day p.o. continuously 7 days per week during concurrent RT (max: 49 days)
  150 mg/M2/day X 5 days; adjuvant cycle #1
  200 mg/M2/day X 5 days; subsequent adjuvant cycles (# 2-12) if tolerability criteria met
  Other Names: Temodar
Procedure: Radiation Therapy — RT will consist of fractionated focal irradiation administered using 2 Gy/fraction, QD x 5 days/week for 6 weeks, for a total dose of 60 Gy

SUMMARY:
Rationale:

In light of the demonstrated activity of anti-angiogenesis agents in rGBM, it is reasonable to postulate that adding these agents to standard RT and chemotherapy in the up-front management of newly diagnosed GBM may improve the clinical benefit. This study will examine the safety and tolerability of adding CT-322 to the standard radiation therapy/temozolomide (RT/TMZ) backbone of treatment for newly diagnosed GBM

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* 18 years or older
* Newly diagnosed, histologically confirmed GBM (grade IV astrocytoma):

  * Subjects will not be eligible if the original histology was a lower grade glioma and a subsequent histological diagnosis of a GBM is made
  * Central independent pathology confirmation of GBM, concurrent with subject enrollment
  * Subjects with sufficient biopsy material available to perform PCR analysis for MGMT promoter methylation must have tissue submitted to the designated laboratory for analysis. Subjects with insufficient tissue or indeterminate results will remain eligible for enrollment.
* KPS ≥ 60
* Be able to begin treatment with RT/TMZ within 6 weeks after biopsy or craniotomy with satisfactory wound healing prior to initiating treatment with CT-322
* Be able to undergo serial MRIs:

  * Measurable or assessable disease may or may not be present
  * CT scanning may not substitute for MRI scanning
* Have adequate bone marrow, liver, renal, and metabolic function as assessed by the following:

  * Hemoglobin ≥ 10.0 g/dL (unsupported)
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3 (unsupported)
  * Platelet count ≥ 100,000/mm3 (unsupported)
  * Total bilirubin ≤ 1.5 x ULN, unless due to Gilbert's disease
  * ALT and AST ≤ 3 x ULN
  * INR < 1.5 or PT within normal limits; and PTT within normal limits
  * Serum creatinine ≤ 1.5 x ULN
  * Urine protein/creatinine ratio (UPCR) < 1.0
  * Serum amylase and lipase ≤ 1.5 x the ULN
* 2-dimensional echo or MUGA scan with LVEF within the institutional normal range
* Stable or decreasing dose of corticosteroids for at least 1 week prior to screening MRI
* Contraceptive measures for male and female participants for the duration of treatment and for 4 weeks following discontinuation of study treatment:

  --Female subjects having reproductive potential must have a negative serum pregnancy test within 72 hours before first administration of CT-322
* Be able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures including receiving daily external beam RT in a radiation treatment facility:

  * integral to or affiliated with the investigative site and in which the treating radiation therapist is a participating study investigator; and
  * that has agreed to follow the radiation treatment guidance and complete the radiation treatment data collection forms

Exclusion Criteria:

* Prior CT-322 therapy or prior therapy with another VEGF-modulating agent (marketed or investigational) for malignant glioma
* History of hypersensitivity to TMZ or any of its excipients, or to Dacarbazine (DTIC)
* Prior treatment for GBM, except surgical resection and/or corticosteroid therapy
* Prior radiotherapeutic, or local (intra-tumoral) or systemic medical therapies (including but not limited to: chemotherapy, hormonal therapy, immunotherapy, anti-angiogenic therapy, implantable Gliadel® wafers, and molecularly targeted therapy) for brain tumors
* Current enrollment in another therapeutic clinical trial involving ongoing therapy
* Concurrent severe and/or uncontrolled medical disease that could compromise participation in the study such as:

  * Pleural or pericardial effusion of ≥ grade 2
  * Uncontrolled diabetes, despite optimal medical management, according to the opinion of the investigator
  * Uncontrolled hypertension (defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management)
  * Any active craniotomy-related wound infection
  * Active clinically significant infection (> grade 2 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events v3.0 (CTCAE) requiring the use of anti-microbial agents, or that would be otherwise, in the opinion of the investigator, interfere with the ability of the subject to participate
  * History of clinically significant bleeding diathesis or coagulopathy including platelet function disorder (e.g., known hemophilia or von Willebrand disease) or acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
  * Ongoing or recent (≤ 3 months) significant gastrointestinal bleeding untreated or recurring
  * Untreated peptic ulcer disease or peptic ulcer disease treated for < 3 months
  * Non-healing wound (including craniotomy wound), ulcer, or bone fracture; or
  * Glomerulonephritis or other protein-wasting glomerulopathy
* Within 12 months before enrollment had:

  * Thrombotic or embolic cerebrovascular accident or transient ischemic attacks
  * CNS bleed (other than stable, grade 1)
  * Intraocular bleed, or any medical condition, which in the opinion of the investigator increases the risk for intra-ocular bleeding
  * Septic endocarditis (unless deemed cured and off all antibiotic therapy for at least 3 months)
  * Coronary artery bypass graft, angioplasty, vascular stenting, myocardial infarction, unstable angina; or
  * Symptomatic congestive heart failure (New York Heart Association ≥ class II)
* Any intraparenchymal CNS hemorrhage at the time of enrollment except for:

  * Grade 1 intraparenchymal hemorrhage in the immediate post-operative period, or
  * Grade 1 intraparenchymal hemorrhage that has been stable (no significant change on 2 consecutive MRI scans at least 4 weeks apart) or improved
* Subjects with a history of prior cardiotoxic chemotherapy exposure or subjects with thoracic irradiation involving cardiac tissue
* Other, non-glioma related major surgery, open biopsy, or significant traumatic injury within 4 weeks before the first dose of CT-322

  --Placement of subcutaneous in-dwelling venous access port within 2 weeks before the first dose of CT-322
* Known human immunodeficiency virus infection or known active acute or chronic viral hepatitis
* Prior malignancy within the previous 3 years, except adequately treated basal cell skin cancer or cervical carcinoma in situ; or if the other primary malignancy is not currently clinically significant or requiring active intervention
* Has any other severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that could increase the risks associated with study participation or study drug administration or could interfere with the interpretation of the study results and, in the judgment of the investigator, would make the subject inappropriate for entry in this study or non-compliant with study-related procedures
* Subjects with medical conditions that would not permit, in the judgment of the investigator, the safe discontinuation of medications that are prohibited throughout the course of the study
* Any condition requiring therapeutic anti-coagulation with either oral (e.g., warfarin type) or injectable anti-coagulants; however, low-dose (i.e., 1 mg daily [QD]) warfarin is permitted for venous port patency maintenance
* Females who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-10 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of CT-322 administered in combination with standard focal brain RT/TMZ to subjects with newly diagnosed GBM | 15 ± 5 days post the last dose of study drug
Establish the recommended Phase 2 dose for the QW schedule of CT-322 for use in this combination | Every 4 weeks until MTD or 2.0 mg/kg dose level is reached

SECONDARY OUTCOMES:
To describe the PK of TMZ and its active metabolite (MTIC) when TMZ is administered alone and when it is co-administered with CT-322 to a subset of approximately 12 subjects with newly diagnosed GBM | Cycle 1, day 1 of RT phase of treatment
To describe the peak and trough concentrations of CT-322 when administered alone and when co-administered with TMZ | RT phase treatment weeks 1-3, 5, 7-10, day 1. Post RT phase cycles 1-3, day 1; then day 1 every 3 cycles thereafter; EOS visit
To evaluate the immunogenicity of CT-322 when administered in combination with standard focal brain RT/TMZ to subjects with newly diagnosed GBM | RT phase treatment weeks 1, 5, 7-8, day 1. Post RT phase cycles 1 and 3, day 1; then day 1 every 3 cycles thereafter; EOS visit
To characterize the plasma biomarker response to CT-322 when administered in combination with standard focal brain RT/TMZ to subjects with newly diagnosed GBM | RT phase treatment weeks 1-3, 5, 7-8, day 1. Post RT phase cycles 1-3, day 1, then day 1 every 3 cycles thereafter; EOS visit

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Kentucky Hospital, Lexington, Kentucky
  - Washington University Cancer Center, St Louis, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina